CLINICAL TRIAL: NCT05793047
Title: Characterization of Fatigue From Data From Inertial Units: Gait Analysis in Hemiplegic Post-stroke Patients
Brief Title: Use of Inertial Sensors to Characterize the Fatigability of Post-stroke Hemiplegic Patients
Acronym: CIMPA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: FondationbHopale (Other)
Responsible Party: Sponsor
Other Study IDs: HOP22-RIPH3-04
Record Dates: First submitted 2023-01-05; First posted 2023-03-31 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Hemiplegic Gait; Fatigue
MeSH Terms: conditions — Gait Disorders, Neurologic; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an experimental, observational, prospective study designed to develop medical knowledge.

The main objective of the study was to identify clinically significant, easily interpretable, quantitative indices of fatigue-related gait pattern changes in post-stroke hemiplegic patients.

This study is part of a usual framework of management of post-stroke hemiplegic patients with additional data collection, via the use of inertial measurement units, considered here as non-interventional.

To achieve this identification, 2 6-minute walk tests will be performed for each patient at the beginning and end of the same day. Patient-perceived fatigue will be recorded by the Borg scale every minute during the 6-minute test. The level of activity during the rehabilitation day is also part of the data collected (number of hours of physical and non-physical activity). At the end of the second 6-minute test, the patient's participation in the study ends.

In addition to the inertial measurement, two scores will be collected to assess the correlation between fatigability and the level of anxiety/depression and stroke severity :

* National Institutes of Health Stroke Scale (NIHSS)
* Hospital Anxiety and Depression Scale (HAD)

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated or entitled to a social security plan
* Patient who has received informed information about the study and who has given his/her consent
* Post-stroke patients (subacute or chronic)
* 1 single unilateral ischemic or hemorrhagic stroke (supratentorial or subtentorial) confirmed by CT or IRM with consecutive hemiparesis
* No lower extremity surgery
* Ability to walk for 6 minutes without human assistance
* Ability to understand instructions in French

Non inclusion Criteria:

* Patients with cognitive problems that prevent them from understanding instructions
* Patent under guardianship or curatorship
* Post-stroke hemiplegic patient (acute = < 6 months)
* Cardiorespiratory pathology incompatible with CT6
* Chronic decompensated pathology
* Neurological pathology
* Orthopedic pathology of the lower limbs or rheumatic conditions that may affect the ability to walk

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients were recruited from among the patients followed for post-stroke rehabilitation at the Jacques Calvé Jacques Calvé rehabilitation center in Berck-sur-Mer.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Relationships between fatigue measured by the Borg scale during 6-minute test and cadence (number of steps per minute) | The 6-minute test takes place at the beginning of the single day of inclusion.Recording of gait characteristics takes place during the entire 6-minute test. The Borg scale will be assessed every minute of the 6-minute test.
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  The Borg Scale is a quantitative measure of perceived exertion during exercise. The Borg scale is rated from 6 to 20. The highest value represents a maximum perception of effort. The Borg scale will be assessed every minute of the 6-minute test.
  Recording of gait characteristics takes place during the entire 6-minute test.
Relationships between fatigue measured by the Borg scale during 6-minute test and walk ratio (stride length / cadence (cm/(steps/min))) | The 6-minute test takes place at the beginning of the single day of inclusion.Recording of gait characteristics takes place during the entire 6-minute test. The Borg scale will be assessed every minute of the 6-minute test.
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  The Borg Scale is a quantitative measure of perceived exertion during exercise. The Borg scale is rated from 6 to 20. The highest value represents a maximum perception of effort. The Borg scale will be assessed every minute of the 6-minute test.
  Recording of gait characteristics takes place during the entire 6-minute test.
Relationships between fatigue measured by the Borg scale during 6-minute test and step length (cm) | The 6-minute test takes place at the beginning of the single day of inclusion.Recording of gait characteristics takes place during the entire 6-minute test. The Borg scale will be assessed every minute of the 6-minute test.
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  The Borg Scale is a quantitative measure of perceived exertion during exercise. The Borg scale is rated from 6 to 20. The highest value represents a maximum perception of effort. The Borg scale will be assessed every minute of the 6-minute test.
  Recording of gait characteristics takes place during the entire 6-minute test.
Relationships between fatigue measured by the Borg scale during 6-minute test and speed (meter per second) | The 6-minute test takes place at the beginning of the single day of inclusion.Recording of gait characteristics takes place during the entire 6-minute test. The Borg scale will be assessed every minute of the 6-minute test.
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  The Borg Scale is a quantitative measure of perceived exertion during exercise. The Borg scale is rated from 6 to 20. The highest value represents a maximum perception of effort. The Borg scale will be assessed every minute of the 6-minute test.
  Recording of gait characteristics takes place during the entire 6-minute test.
Relationships between fatigue measured by the Borg scale during 6-minute test and cycles phases: single and double support (second) | The 6-minute test takes place at the beginning of the single day of inclusion.Recording of gait characteristics takes place during the entire 6-minute test. The Borg scale will be assessed every minute of the 6-minute test.
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  The Borg Scale is a quantitative measure of perceived exertion during exercise. The Borg scale is rated from 6 to 20. The highest value represents a maximum perception of effort. The Borg scale will be assessed every minute of the 6-minute test.
  Recording of gait characteristics takes place during the entire 6-minute test.
Relationships between fatigue measured by the Borg scale during 6-minute test and postural control: step width (cm) and standard deviation (cm) | The 6-minute test takes place at the beginning of the single day of inclusion.Recording of gait characteristics takes place during the entire 6-minute test. The Borg scale will be assessed every minute of the 6-minute test.
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  The Borg Scale is a quantitative measure of perceived exertion during exercise. The Borg scale is rated from 6 to 20. The highest value represents a maximum perception of effort. The Borg scale will be assessed every minute of the 6-minute test.
  Recording of gait characteristics takes place during the entire 6-minute test.
Relationships between fatigue measured by the Borg scale during 6-minute test and asymmetry dtermined by stride length ratio and single stance duration ratio | The 6-minute test takes place at the beginning of the single day of inclusion.Recording of gait characteristics takes place during the entire 6-minute test. The Borg scale will be assessed every minute of the 6-minute test.
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  The Borg Scale is a quantitative measure of perceived exertion during exercise. The Borg scale is rated from 6 to 20. The highest value represents a maximum perception of effort. The Borg scale will be assessed every minute of the 6-minute test.
  Recording of gait characteristics takes place during the entire 6-minute test.
Relationships between fatigue measured by the Borg scale during 6-minute test and cadence (number of steps per minute) | The 6-minute test takes place at the end of the single day of inclusion.Recording of gait characteristics takes place during the entire 6-minute test. The Borg scale will be assessed every minute of the 6-minute test.
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  The Borg Scale is a quantitative measure of perceived exertion during exercise. The Borg scale is rated from 6 to 20. The highest value represents a maximum perception of effort. The Borg scale will be assessed every minute of the 6-minute test.
  Recording of gait characteristics takes place during the entire 6-minute test.
Relationships between fatigue measured by the Borg scale during 6-minute test and walk ratio (stride length / cadence (cm/(steps/min))) | The 6-minute test takes place at the end of the single day of inclusion.Recording of gait characteristics takes place during the entire 6-minute test. The Borg scale will be assessed every minute of the 6-minute test.
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  The Borg Scale is a quantitative measure of perceived exertion during exercise. The Borg scale is rated from 6 to 20. The highest value represents a maximum perception of effort. The Borg scale will be assessed every minute of the 6-minute test.
  Recording of gait characteristics takes place during the entire 6-minute test.
Relationships between fatigue measured by the Borg scale during 6-minute test and step length (cm) | The 6-minute test takes place at the end of the single day of inclusion.Recording of gait characteristics takes place during the entire 6-minute test. The Borg scale will be assessed every minute of the 6-minute test
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  The Borg Scale is a quantitative measure of perceived exertion during exercise. The Borg scale is rated from 6 to 20. The highest value represents a maximum perception of effort. The Borg scale will be assessed every minute of the 6-minute test.
  Recording of gait characteristics takes place during the entire 6-minute test.
Relationships between fatigue measured by the Borg scale during 6-minute test and speed (meter per second) | The 6-minute test takes place at the end of the single day of inclusion.Recording of gait characteristics takes place during the entire 6-minute test. The Borg scale will be assessed every minute of the 6-minute test.
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  The Borg Scale is a quantitative measure of perceived exertion during exercise. The Borg scale is rated from 6 to 20. The highest value represents a maximum perception of effort. The Borg scale will be assessed every minute of the 6-minute test.
  Recording of gait characteristics takes place during the entire 6-minute test.
Relationships between fatigue measured by the Borg scale during 6-minute test and cycles phases: single and double support (second) | The 6-minute test takes place at the end of the single day of inclusion.Recording of gait characteristics takes place during the entire 6-minute test. The Borg scale will be assessed every minute of the 6-minute test.
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  The Borg Scale is a quantitative measure of perceived exertion during exercise. The Borg scale is rated from 6 to 20. The highest value represents a maximum perception of effort. The Borg scale will be assessed every minute of the 6-minute test.
  Recording of gait characteristics takes place during the entire 6-minute test.
Relationships between fatigue measured by the Borg scale during 6-minute test and postural control: step width (cm) and standard deviation (cm) | The 6-minute test takes place at the end of the single day of inclusion.Recording of gait characteristics takes place during the entire 6-minute test. The Borg scale will be assessed every minute of the 6-minute test.
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  The Borg Scale is a quantitative measure of perceived exertion during exercise. The Borg scale is rated from 6 to 20. The highest value represents a maximum perception of effort. The Borg scale will be assessed every minute of the 6-minute test.
  Recording of gait characteristics takes place during the entire 6-minute test.
Relationships between fatigue measured by the Borg scale during 6-minute test and asymmetry determined by stride length ratio and single stance duration ratio | The 6-minute test takes place at the end of the single day of inclusion.Recording of gait characteristics takes place during the entire 6-minute test. The Borg scale will be assessed every minute of the 6-minute test.
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  The Borg Scale is a quantitative measure of perceived exertion during exercise. The Borg scale is rated from 6 to 20. The highest value represents a maximum perception of effort. The Borg scale will be assessed every minute of the 6-minute test.
  Recording of gait characteristics takes place during the entire 6-minute test.
Change cadence (number of steps per minute) in fonction of the fatigue measured by the Borg scale recorded during the two 6-minute tests | Change of the gait parameter between the beginning of the single day of inclusion (before the rehabilitation) and the end of the single day of inclusion (after the rehabilitation sessions).
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  The Borg Scale is a quantitative measure of perceived exertion during exercise. The Borg scale is rated from 6 to 20. The highest value represents a maximum perception of effort. The Borg scale will be assessed every minute of the 6-minute test.
  Recording of gait characteristics takes place during the entire 6-minute test.
Change walk ratio (stride length / cadence (cm/(steps/min))) in fonction of the fatigue measured by the Borg scale recorded during the two 6-minute tests | Change of the gait parameter between the beginning of the single day of inclusion (before the rehabilitation) and the end of the single day of inclusion (after the rehabilitation sessions).
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  The Borg Scale is a quantitative measure of perceived exertion during exercise. The Borg scale is rated from 6 to 20. The highest value represents a maximum perception of effort. The Borg scale will be assessed every minute of the 6-minute test.
  Recording of gait characteristics takes place during the entire 6-minute test.
Change step length (cm) in fonction of the fatigue measured by the Borg scale recorded during the two 6-minute tests | Change of the gait parameter between the beginning of the single day of inclusion (before the rehabilitation) and the end of the single day of inclusion (after the rehabilitation sessions).
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  The Borg Scale is a quantitative measure of perceived exertion during exercise. The Borg scale is rated from 6 to 20. The highest value represents a maximum perception of effort. The Borg scale will be assessed every minute of the 6-minute test.
  Recording of gait characteristics takes place during the entire 6-minute test.
Change speed (meter per second) in fonction of the fatigue measured by the Borg scale recorded during the two 6-minute tests | Change of the gait parameter between the beginning of the single day of inclusion (before the rehabilitation) and the end of the single day of inclusion (after the rehabilitation sessions).
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  The Borg Scale is a quantitative measure of perceived exertion during exercise. The Borg scale is rated from 6 to 20. The highest value represents a maximum perception of effort. The Borg scale will be assessed every minute of the 6-minute test.
  Recording of gait characteristics takes place during the entire 6-minute test.
Change cycle phase: single and double support (second) in fonction of the fatigue measured by the Borg scale recorded during the two 6-minute tests | Change of the gait parameter between the beginning of the single day of inclusion (before the rehabilitation) and the end of the single day of inclusion (after the rehabilitation sessions).
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  The Borg Scale is a quantitative measure of perceived exertion during exercise. The Borg scale is rated from 6 to 20. The highest value represents a maximum perception of effort. The Borg scale will be assessed every minute of the 6-minute test.
  Recording of gait characteristics takes place during the entire 6-minute test.
Change postural control: step width (cm) and standard deviation (cm) in fonction of the fatigue measured by the Borg scale recorded during the two 6-minute tests | Change of the gait parameter between the beginning of the single day of inclusion (before the rehabilitation) and the end of the single day of inclusion (after the rehabilitation sessions).
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  The Borg Scale is a quantitative measure of perceived exertion during exercise. The Borg scale is rated from 6 to 20. The highest value represents a maximum perception of effort. The Borg scale will be assessed every minute of the 6-minute test.
  Recording of gait characteristics takes place during the entire 6-minute test.
Change asymmetry: stride length ratio; single stance duration ratio in fonction of the fatigue measured by the Borg scale recorded during the two 6-minute tests | Change of the gait parameter between the beginning of the single day of inclusion (before the rehabilitation) and the end of the single day of inclusion (after the rehabilitation sessions).
  The 6-min walk test (TM6) measures the greatest distance covered in 6 min of walking around two studs separated by 30 meters.
  The Borg Scale is a quantitative measure of perceived exertion during exercise. The Borg scale is rated from 6 to 20. The highest value represents a maximum perception of effort. The Borg scale will be assessed every minute of the 6-minute test.
  Recording of gait characteristics takes place during the entire 6-minute test.

SECONDARY OUTCOMES:
To assess the correlation between fatigability and the level of anxiety/depression | During the one day of patient assessment. Assessed only once for each patient before performing the first 6-minute test.
  Questionnaire Hospital Anxiety and Depression scale (HAD) The Hospital Anxiety and Depression scale (HAD) questionnaire is used to screen for anxiety and depressive disorders. It includes 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), thus making it possible to obtain two scores (maximum score for each score: 21). A score close to 0 means no anxiety symptoms a score close to 11 and above indicates anxiety symptoms. This scale is validated in French.
To assess the correlation between fatigability and stroke severity | During the one day of patient assessment. Assessed only once for each patient before performing the first 6-minute test.
  National Institutes of Health Stroke Scale (NIHSS) The National Institutes of Health Stroke Scale (NIHSS) is a 15-item impairment rating scale designed to assess the neurological consequences and degree of recovery of a stroke patient.
  Total scores on the NIHSS range from 0 to 42, with higher values reflecting more severe brain damage.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal RIGAUX, Principal Investigator — Hopale Foundation - Jacques Calvé Institute
Locations (1):
- Institut Calvé, Berck, France

IPD SHARING:
Plan to Share IPD: No